CLINICAL TRIAL: NCT00242996
Title: Phase II Trial of Rituximab and Autologous Stem Cell Transplantation for Refractory B Cell Large Cell Lymphoma
Brief Title: Rituximab, Cyclophosphamide, and G-CSF Followed By Combination Chemotherapy in Treating Patients Who Are Undergoing Autologous Stem Cell Transplant Followed By Rituximab and GM-CSF for Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: J0376 CDR0000447158; P30CA006973 (NIH); JHOC-J0376; WIRB-20040009
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Rituximab; sargramostim; Carmustine; Cyclophosphamide; Etoposide; Chemotherapy, Adjuvant; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Biological: sargramostim
Drug: carmustine
Drug: cyclophosphamide
Drug: etoposide
Procedure: adjuvant therapy
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving colony-stimulating factors, such as G-CSF, monoclonal antibodies, such as rituximab, and chemotherapy, such as cyclophosphamide, helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored for peripheral stem cell transplant. Giving chemotherapy, such as carmustine, etoposide, and cyclophosphamide, before transplant stops the growth of cancer cells by stopping them from dividing or killing them. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. More rituximab is given after transplant to kill any remaining cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with cyclophosphamide and G-CSF followed by combination chemotherapy works in treating patients undergoing an autologous stem cell transplant followed by rituximab and GM-CSF for refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the disease-free and overall survival of patients with refractory diffuse large B-cell lymphoma treated with stem cell mobilization comprising rituximab, cyclophosphamide, and filgrastim (G-CSF) followed by high-dose chemotherapy comprising carmustine, etoposide, and cyclophosphamide and autologous peripheral blood stem cell transplantation, rituximab, and sargramostim (GM-CSF).
* Determine any potential infectious complications in patients treated with this regimen.
* Determine the effect of GM-CSF on antibody-dependent cellular cytotoxicity in patients treated with this regimen.

OUTLINE: Stem cell mobilization: Patients receive rituximab IV over 4-8 hours on days 1, 5, 8, and 13. Patients also receive cyclophosphamide IV over 1-2 hours on day 9 and filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 10 and continuing until an adequate number of peripheral blood stem cells (PBSC) are collected.

High-dose preparative regimen: Patients receive carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 2 hours on day -2.

Autologous PBSC transplantation: Patients undergo autologous PBSC transplantation on day 0. Patients receive sargramostim (GM-CSF) SC once daily beginning on day 6 and continuing until blood counts recover.

Post-transplant regimen: Patients receive GM-CSF SC once daily on days 42-73, 177-208, 362-393, 543-574, and 727-758. Patients also receive rituximab IV over 4-8 hours on days 45, 52, 59, 66, 180,187, 194, 201, 365, 372, 379, 386, 546, 553, 560, 567, 730, 737, 744, and 751.

After completion of study treatment, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell lymphoma, meeting 1 of the following criteria:

  * Failed to achieve at least partial remission
  * Failed to respond to prior primary therapy or salvage chemotherapy
  * Disease progression within 6 weeks after achieving remission
* CD20 expression at diagnosis or relapse
* No more than 4 prior regimens using chemotherapy, radiotherapy, or immunotherapy

  * The addition of radiotherapy or a monoclonal antibody to chemotherapy is considered 1 treatment regimen provided the addition was part of the initial treatment plan

    * The addition of these therapies due to lack of response or poor response is considered an additional treatment regimen whether given in the front line or salvage setting

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Direct bilirubin ≤ 2 mg/dL
* AST or ALT < 3 times upper limit of normal

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* Ejection fraction ≥ 40%

Pulmonary

* DLCO ≥ 60% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 2 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No active infection requiring oral or IV antibiotics
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Radiotherapy

Chemotherapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* No prior radioimmunotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
2-year event free survival

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States